CLINICAL TRIAL: NCT05319067
Title: Study of Gut Microbiota Diversity in Children Aged 1-3 Years on Prolonged Antibiotic Prophylaxis for Grade 3 or Higher Vesicoureteral Reflux Compared With 2 Age-matched Control Groups
Acronym: PROPHYBIOTA
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: NIMAO/2021-2/AF-01
Record Dates: First submitted 2022-04-01; First posted 2022-04-08 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Vesicoureteral Reflux 3
Keywords: Antibiotic prophylaxis; Microbiota

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cases: Children aged 1 to 3 years with vesico ureteral reflux of grade 3 or higher, under antibiotic prophylaxis
  Interventions: Other: Stool sampling
- Controls: Children aged 1 to 3 years with uropathy, without antibiotic prophylaxis
  Interventions: Other: Stool sampling
- Healthy Controls: Healthy children aged 1 to 3 years.
  Interventions: Other: Stool sampling

INTERVENTIONS:
Other: Stool sampling — Stool sample taken at home 24 hours before hospital visit

SUMMARY:
Urinary tract infections are very common in pediatrics. Urinary antibiotic prophylaxis is commonly used in children with malformative uropathies. Long-term, low-dose antibiotic prophylaxis with trimethoprim-sulfamethoxazole has been associated with a decrease in the number of urinary tract infections in susceptible children, but not systematically with a decrease in the risk of renal scarring (depending of uropathy stage).

Long-term antibiotic prophylaxis has implications for the acquisition of antibiotic resistance. A child receiving antibiotic prophylaxis for urinary tract infection is around 6 times more likely to develop a multidrug-resistant infection. In the general population, the microbiota of children treated with curative antibiotics is less diverse in terms of species and strains. In addition, short-term compositional changes are observed between consecutive samples of children treated with antibiotics.

The gut microbiota modulates the immune system, in particular via metabolites (SCFA, polysaccharide A) produced by bacteria that modify the expansion and function of regulatory T-cells. The disturbances of the intestinal microbiota play a role in the medium and long term on the acquisition of pathologies, such as atopy.

The study authors wish to describe the intestinal microbiota of children with vesico-ureteral reflux treated long-term with trimethoprim-sulfamethoxazole and compared it those not receiving antibiotic prophylaxis and to healthy children.

ELIGIBILITY:
Inclusion Criteria:

* The patient must be a member or beneficiary of a health insurance plan
* Patient with no objection to participation in the study from the parent or guardian
* Child with a diversified diet.

  o Specific inclusion criteria for group 1 (cases):
* Child with grade 3 or higher vesicoureteral reflux.
* Child on trimethoprim-sulfamethoxazole therapy for at least 5 months.

  o Specific inclusion criteria for group 2 (controls):
* Child with uropathy and without long-term trimethoprim-sulfamethoxazole treatment.

  o Specific inclusion criteria for group 3 (healthy controls):
* Child without uropathy or long-term trimethoprim-sulfamethoxazole treatment.

Exclusion Criteria:

* Chronic digestive pathology
* Acute gastroenteritis or infectious colitis within last 15 days.
* Curative antibiotic therapy taken less than one month ago.
* Chronic inflammatory bowel disease or other localizations
* Congenital or acquired immune deficiency (current treatment with methotrexate, biotherapies, immunosuppressants)
* Patient participating in a category 1 trial likely to modify the intestinal microbiota.
* Patient in an exclusion period determined by another study.
* Patient under court protection, guardianship or curatorship.
* Patient for whom it is impossible to give informed information to person with parental authority.

Ages: 1 Year to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: For the purpose of the study three groups of children will be constituted:
  Children aged 1 to 3 years with vesico ureteral reflux of grade 3 or higher, under antibiotic prophylaxis; Children aged 1 to 3 years with uropathy, without antibiotic prophylaxis; Controls: Healthy children aged 1 to 3 years.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
α-diversity of the gut microbiota between groups | Day 0
  N index of a stool sample measured by the Shannon index (H^') which incorporates the total number of different Operational Taxonomic Units and the relative proportions of these Operational Taxonomic Units.

SECONDARY OUTCOMES:
The β-diversity of the gut microbiota between groups | Day 0
  Operational Taxonomic Units measured by Bray Curtis Index
The number of bacterial genera present in the gut microbiota between groups | Day 0
  Relative abundance Operational Taxonomic Units present
The prevalence of multi-resistant bacteria | Day 0
  % of isolated bacteria producing extended spectrum betalactamase, carbapenemase-producing Enterococcus faecium and glycopeptide-resistant Enterococcus faecium and bacteria resistant to trimethoprim-sulfamethoxazole

CONTACTS AND LOCATIONS:
Overall Officials: Anne Filleron, Principal Investigator — CHU de Nimes
Locations (2):
- France (2):
  - CHU de Montpellier, Montpellier
  - CHU de Nîmes, Nîmes